CLINICAL TRIAL: NCT01099527
Title: A Phase I/II Trial of RAD001/Capecitabine in Refractory Gastric Cancer
Brief Title: A Trial of RAD001/Capecitabine in Refractory Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Samsung Medical center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-02-041
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Metastatic Gastric Cancer
Keywords: gastric cancer; refractory; metastatic
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Everolimus; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental): Everolimus (RAD001) dose escalation of capecitabine, everolimus
  Capecitabine dose escalation of capecitabine, everolimus
  Interventions: Drug: Everolimus (RAD001); Drug: Capecitabine

INTERVENTIONS:
Drug: Everolimus (RAD001) — dose escalation of capecitabine, everolimus
Drug: Capecitabine — dose escalation of capecitabine, everolimus

SUMMARY:
Capecitabine is an oral fluoropyrimidine that has been shown to be effective in the treatment of metastatic gastric and colorectal cancer patients. On the basis of capecitabine-based chemotherapy which is accepted as a standard regimen in gastric cancer, we will perform the phase I/II study with all-oral regimen of RAD001 with capecitabine for these refractory gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven gastric cancer patients
2. Adequate organ function as defined by the following criteria:

   A. Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase (SGOT)) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase (SGPT)) ≤ 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy B. Total serum bilirubin ≤ 3.0 mg/dL C. Absolute neutrophil count (ANC) ≥1500/µL D. Platelets ≥100,000/µL E. Hemoglobin ≥9.0 g/dL (may be transfused or erythropoietin treated) F. Serum calcium ≤12.0 mg/dL G. Serum creatinine ≤1.5 x ULN
3. Patients with CNS metastasis must have stable neurologic function without evidence of CNS progression within 8 weeks
4. Patients who have failed to at least two previous cytotoxic chemotherapy for advanced gastric cancer (adjuvant treatment will be counted as one regimen if received < 12 months from the start of experimental treatment)
5. At least one measurable lesion by RECIST criteria
6. ECOG PS 0-2
7. Patients with informed consent

Exclusion Criteria:

1. Major surgery or radiation therapy within 4 weeks of starting the study treatment.
2. History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease on screening CT or MRI scan.
3. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2.
4. Pregnancy or breastfeeding.
5. Prior exposure to the study drug.
6. Patients unable to swallow oral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-10; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine maximum tolerated dose (MTD) in phase I | 1 year
To assess response rate in phase II | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Cancer Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee SJ, Lee J, Lee J, Park SH, Park JO, Park YS, Lim HY, Kim KM, Do IG, Jung SH, Yim DS, Kang WK. Phase II trial of capecitabine and everolimus (RAD001) combination in refractory gastric cancer patients. Invest New Drugs. 2013 Dec;31(6):1580-6. doi: 10.1007/s10637-013-0022-0. Epub 2013 Sep 7. PMID 24013904